CLINICAL TRIAL: NCT00329654
Title: A Prospective, Randomized, Single Blinded, Controlled Clinical Investigation of James Embar® Light Therapy in the Treatment of Burn Wounds With Little Healing Potential
Brief Title: James EMBAR® Light Therapy in the Treatment of Burn Wounds of Intermediate Depth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Tendris Holding BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2006/067
Record Dates: First submitted 2006-05-23; First posted 2006-05-25 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Burns
Keywords: Burn wounds, light therapy
MeSH Terms: conditions — Burns | interventions — Phototherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Embar® light therapy or sham irradiation (Experimental): Phototherapy with the Embar® light therapy or sham irradiation.
  Interventions: Procedure: Phototherapy with the Embar® light therapy or sham irradiation

INTERVENTIONS:
Procedure: Phototherapy with the Embar® light therapy or sham irradiation — Phototherapy with the Embar® light therapy or sham irradiation is followed.

SUMMARY:
This will be a prospective, randomized, single blinded, controlled study in a single center setting to assess the effect of either phototherapy with the Embar® light therapy or sham irradiation.

DETAILED DESCRIPTION:
This will be a prospective, randomized, single blinded, controlled study in a single center setting. Patients with burn wounds will be screened for enrollment. All burn wounds that are not clearly full thickness on clinical assessment will be treated the first 48 to 72 hours with a hydrocolloid gel (Flaminal®) combined with Vaseline gauze. Wounds will be photographed on a daily basis. In order to obtain an optimal preparation for Laser Doppler imaging, the burn wounds will be meticulously debrided during dressing changes. Patients whose burn wound meet the inclusion criteria will be randomized to receive either phototherapy with the Embar® light therapy or sham irradiation. Disinfection and topical treatment of the wounds will be the same in both groups as well as the treatment regimen after wound closure with special pressure garments and hydration.

Clinical wound assessments, wound tracings (if possible) and digital photographs will be conducted at least twice a week till wound healing. Swabs will be taken on admission, the day after laser Doppler imaging and from then on a weekly basis. Primary endpoint is complete epithelialization of the wound, secondary endpoint is maturation of the scar after one year. Follow-Ups will be performed one, three, six and twelve months after wound closure. The treatment regimen will consist of custom made pressure garments and hydration of the scar. Objective methods will be used during these follow-ups to evaluate elasticity and color of the scar, this by using the Dermalab and the Dermaspectrometer, as well as the Vancouver Scar Scale, a subjective method.

ELIGIBILITY:
Inclusion Criteria:

* All burn wounds with flux values measured by Laser Doppler Imaging, corresponding with expected healing time between 14 and 21 days, flux values between 200 and 600 (Pink-Yellow-Green-Light Blue color)
* All burn wounds with above mentioned values and a maximal size of 8 by 10 cm.
* Wounds treated with a hydrocolloid gel prior to LDI
* All assessments are done during first days before scanning
* Patients wish and possibility to follow the complete treatment schedule till wound healing and participation on complete follow-up schedule
* Informed consent has been obtained

Exclusion Criteria:

* All burn wounds with flux values measured by Laser Doppler Imaging, corresponding with other healing times (Red and Dark blue color)
* Impossibility to debride necrotic skin prior to LDI measurement
* All burn wounds with values for inclusion but above the maximal wound size
* Wounds treated with other topical ointments than hydrocolloids
* Not following the complete treatment schedule or missing some evaluations during the follow-up period
* Patient has any condition(s) that seriously compromises the patient's ability to complete this study.
* Patient has participated in another study utilizing an investigational drug or device within the previous 30 days
* Patient has one or more medical condition(s), diabetes, including renal, hepatic, hematologic, neurologic, or immune disease that in the opinion of the investigator would make the patient an inappropriate candidate for this wound healing study
* The plastic surgeon decides that surgery is necessary
* Patients wish to terminate the study
* No informed consent before start of the trial

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Wound closure | At time T0

SECONDARY OUTCOMES:
Scar assessment | 1 month, 3 months, 6 months and 1 year after wound closure
  Scar assessment will be followed

CONTACTS AND LOCATIONS:
Overall Officials: Stan Monstrey, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be